CLINICAL TRIAL: NCT06951633
Title: Functional Efficiency, Respiratory Parameters and Blood Rheological Tests in Elderly People With Respiratory Diseases Participating in Pulmonary Rehabilitation in Underground Salt Chambers - a Prospective Experimental Study, Controlled in a Crossover Design
Brief Title: Effects of Pulmonary Rehabilitation in Salt Chambers on Functional Efficiency, Respiratory Parameters, and Blood Rheology in Elderly With Respiratory Diseases.
Acronym: PRSC-FERPBR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University School of Physical Education, Krakow, Poland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 29/RID/2025; No. 022/ RID/SP/0027/2024/01 (Other Grant/Funding Number: Minister of Science and Higher Education)
Record Dates: First submitted 2025-04-07; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: the Elderly; Respiratory Disorders
Keywords: Pulmonary function, speleotherapy, blood tests, 6MWT, chest
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Intervention Model Description: A Prospective, Controlled, Crossover Study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Subterranean, pulmonary rehabilitation (Other): Pulmonary rehabilitation in the underground salt chambers of the 'Wieliczka' Salt Mine Health Resort
  Interventions: Other: Subterranean, pulmonary rehabilitation

INTERVENTIONS:
Other: Subterranean, pulmonary rehabilitation — Pulmonary rehabilitation in the underground Health Resort of the 'Wieliczka' Salt Mine

SUMMARY:
The aim of the study is to assess the impact of the rehabilitation and treatment stay at the underground Health Resort of the 'Wieliczka' Salt Mine in Wieliczka on the functional capacity, respiratory parameters, and rheological properties of blood in elderly individuals with respiratory diseases.

DETAILED DESCRIPTION:
The research project will involve patients aged 65 and older with chronic respiratory diseases. Based on controlled studies conducted at the Health Resort "Wieliczka" Salt Mine in Wieliczka, and assuming the project will be a prospective, experimental, controlled study with a crossover design, calculations were made for the primary variable under investigation (exercise tolerance). These calculations determined that 29 pairs of participants are needed to achieve a statistical power of 80% and a significance level of 5% (bilateral). To detect a mean difference between pairs of 58, assuming a standard deviation of 106 for these differences and accounting for a 10% loss of participants from observation, the required sample size was increased to 33 pairs. Given the crossover design, the study plans to include 33 patients.

Volunteers will undergo qualifying tests, measurements of functional fitness, respiratory indicators, and blood rheology tests 3 weeks prior to the start of the rehabilitation and therapeutic stay in the underground salt chambers (1st test). During the 3-week period before the rehabilitation, participants will not engage in any other form of therapeutic rehabilitation. Functional fitness, respiratory indicators, and blood rheology tests will be repeated before the start of the stay (2nd test), immediately after its completion (3rd test), and 3 months after its completion (4th follow-up test). Each day of the rehabilitation and therapeutic stay will include a 2.5-hour visit to the underground health resort under the supervision of a doctor, physiotherapist, and nurse, during which pulmonary rehabilitation will be implemented.

ELIGIBILITY:
Inclusion Criteria:

* people aged 65 and older with chronic respiratory diseases in a stable period of the disease (without exacerbations), qualified to participate in a rehabilitation and treatment stay in the underground Health Resort 'Wieliczka' Salt Mine in Wieliczka,
* patients who gave informed, written consent to participate in the study.

Exclusion Criteria:

* patients with contraindications to subterraneotherapy and physical exercise,
* lack of written consent to participate in the study,
* deterioration of health during the implementation of the program.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-04-04 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Respiratory muscle force: Maximal inspiratory pressure - MIP | up to 18 months
  This test involves wearing a nose peg and inhaling through a tube, performed in three trials.
Respiratory muscle force: Maximal expiratory pressure - MEP | up to 18 months
  This test involves wearing a nose peg and exhaling through a tube, performed in three trials.
Respiratory muscle force: Sniff Nasal Inspiratory Pressure - SNIP | up to 18 months
  The test consists of separate inhalations through the left and right nostrils, performed in five trials per nostril.
6-Minute Walk Test - 6MWT | up to 18 months
  The 6-Minute Walk Test (6MWT) is a standardized test used to assess functional exercise capacity. It measures the distance an individual can walk on a flat, hard surface in a period of six minutes
The Aggregation Index (AI) | up to 18 months
  The Aggregation Index (AI), indicating the extent of red blood cell aggregation, is measured using the Lorrca Maxis (Laser-Assisted Optical Rotational Cell Analyzer) under standardized shear conditions.
  (AI) analyzed
The half-time of total aggregation (T1/2) | up to 18 months
  The half-time of total aggregation (T1/2), which reflects the time required for red blood cells to aggregate to 50% of their maximum value, is assessed using the Lorrca Maxis (Laser-Assisted Optical Rotational Cell Analyzer). This test measures the aggregation kinetics of erythrocytes under controlled shear stress, providing a quantitative assessment of the aggregation process.
The Elongation Index (EI) | up to 18 months
  The Elongation Index (EI), reflecting red blood cell deformability, is measured using the Lorrca Maxis (Laser-Assisted Optical Rotational Cell Analyzer), which evaluates the ability of erythrocytes to deform under varying shear stress.
4- Meters Gait Speed Test - 4MGST | up to 18 months
  The 4-Meters Gait Speed Test (4MGST) is a simple, widely used assessment tool to measure an individual's walking speed over a short, fixed distance. It is primarily used to evaluate mobility and functional performance, especially in elderly individuals.
Health Related Quality of Life - HRQoL withe the use of 15D questionnaire. | up to 18 months
  The 15D is a comprehensive, generic health-related quality of life (HRQoL) tool that measures an individual's overall health status. It includes 15 dimensions, covering aspects of physical, mental, and social well-being.Minimum Value: 0 (representing the worst possible health state)
  Maximum Value: 1 (representing the best possible health state). Higher Scores indicate better health-related quality of life, reflecting higher levels of functioning and well-being across the 15 dimensions.
Chest mobility | up to 18 months
  The assessment of chest mobility involves evaluating the range of motion (ROM) and the expansion of the chest during inspiration and expiration, performed in three trials.
Back scratch test | up to 18 months
  The patient is instructed to reach with his dominant hand behind his head, over the shoulder, as if trying to scratch the back of their neck. The fingers should be pointing downward toward the spine.The distance between the fingers (or whether they touch) is measured to assess the flexibility and range of motion of the shoulder and upper back.
Interleukin IL 1b | up to 18 months
  Interleukin-1 beta (IL-1β) is a pro-inflammatory cytokine produced primarily by activated macrophages and monocytes. It plays a central role in the regulation of immune and inflammatory responses and is considered a key mediator in the pathophysiology of various chronic inflammatory, autoimmune, and infectious diseases.
Interleukin IL-6 | up to 18 months
  Interleukin-6 (IL-6) is a pleiotropic pro-inflammatory cytokine produced by various cell types, including macrophages, T cells, B cells, endothelial cells, fibroblasts, and skeletal muscle cells. It plays a key role in the regulation of immune responses, inflammation, hematopoiesis, and metabolism.
TNF-alfa | up to 18 months
  Tumor Necrosis Factor alpha (TNF-α) is a key pro-inflammatory cytokine involved in the regulation of immune responses, inflammation, and apoptosis. It is produced primarily by activated macrophages, but also by T lymphocytes, natural killer (NK) cells, and other immune and non-immune cells in response to infection, injury, or immune stimulation.
WBC [10⁹/l] | up to 18 months
  White Blood Cell Count - WBC [10⁹/l]
  Represents the number of leukocytes in one liter of blood. WBCs play a crucial role in immune defense. Elevated levels may indicate infection, inflammation, physiological stress, or hematologic malignancies. Decreased levels can be associated with bone marrow suppression or immunodeficiency.
RBC [10¹²/l], | up to 18 months
  Red Blood Cell Count - RBC [10¹²/l]
  Indicates the number of erythrocytes per liter of blood. RBCs are responsible for oxygen transport. Decreased levels suggest anemia; elevated levels may indicate dehydration or polycythemia.
HGB [g/dl] | up to 18 months
  Hemoglobin Concentration - HGB [g/dl]
  Measures the amount of hemoglobin in the blood. Hemoglobin is the oxygen-carrying protein in red blood cells. It is a key indicator of oxygen-carrying capacity and a primary marker for diagnosing anemia.
HCT [%] | up to 18 months
  Hematocrit - HCT [%]
  Refers to the percentage of total blood volume occupied by red blood cells. Lower values are commonly seen in anemia; higher values may indicate dehydration or polycythemia.
MCV [fl] | up to 18 months
  Mean Corpuscular Volume - MCV [fl]
  Reflects the average volume of individual erythrocytes. It helps to classify anemia as microcytic, normocytic, or macrocytic.
MCH [pg] | up to 18 months
  Mean Corpuscular Hemoglobin -MCH [pg]
  Indicates the average amount of hemoglobin per red blood cell. It provides additional insight into the hemoglobin content in different types of anemia.
MCHC [g/dl] | up to 18 months
  Mean Corpuscular Hemoglobin Concentration - MCHC [g/dl]
  Represents the average concentration of hemoglobin in erythrocytes. Decreased levels suggest hypochromia, commonly observed in iron deficiency anemia.
PLT [109/l] | up to 18 months
  Platelet Count - PLT [10⁹/l]
  Determines the number of platelets in one liter of blood. Platelets are essential for blood clotting. Thrombocytopenia increases bleeding risk, while elevated platelet counts may indicate inflammation or a prothrombotic state.
Reticulocytes {% or ‰] | up to 18 months
  Reticulocytes [% or ‰]
  Immature red blood cells that reflect bone marrow erythropoietic activity. Increased reticulocyte counts indicate active regeneration, commonly seen in response to anemia or blood loss.
CRP [mg/l] | up to 18 months
  C-Reactive Protein - CRP [mg/l]
  An acute-phase protein produced by the liver in response to inflammation. Elevated CRP levels are a sensitive but non-specific marker of acute inflammation, infection, or tissue injury.
Fibrinogen [g/l] | up to 18 months
  Fibrinogen
  A coagulation factor and acute-phase reactant synthesized in the liver. Increased fibrinogen levels are observed during inflammation, infection, or trauma and may contribute to a hypercoagulable state.
ESR [mm/h] | up to 18 months
  Erythrocyte Sedimentation Rate - ESR [mm/h]
  A non-specific indicator of inflammation that measures the rate at which red blood cells settle in a vertical tube over one hour. Elevated ESR values are commonly found in infections, autoimmune diseases, and malignancies.

SECONDARY OUTCOMES:
FEV₁ | 2 weeks
  Forced Expiratory Volume in One Second [L] - FEV₁
  FEV₁ represents the volume of air forcibly exhaled during the first second of a forced expiratory maneuver, starting from full lung inflation.
  It is a key parameter in the assessment of airway obstruction and is used in the diagnosis and monitoring of diseases such as chronic obstructive pulmonary disease (COPD) and asthma.
  Lower FEV₁ values indicate narrowing of the airways or reduced lung function.
FVC | 2 weeks
  Forced Vital Capacity [L] - FVC
  FVC is the total volume of air that can be forcibly exhaled after a full inspiration.
  It reflects the elastic properties of the lungs and chest wall. FVC is used in conjunction with FEV₁ to assess restrictive and obstructive ventilatory patterns. A reduced FVC may suggest lung restriction, while a low FEV₁/FVC ratio typically indicates airway obstruction.
PEF | 2 weeks
  Peak Expiratory Flow [L/min] - PEF
  PEF represents the maximum flow rate achieved during a forced expiratory maneuver.
  It is a simple and reproducible indicator of large airway function and is often used in asthma monitoring, bronchodilator response testing, and occupational lung health assessments.
  Reduced PEF may indicate airway narrowing, poor effort, or respiratory muscle weakness.
Bronchodilator Reversibility (BDR) Test | 2 weeks
  The bronchodilator reversibility test is performed to assess the responsiveness of the airways to bronchodilator medications, typically in patients suspected of having reversible airway obstruction, such as in asthma or chronic obstructive pulmonary disease (COPD).
  The test evaluates how spirometric values change following the administration of a bronchodilator (e.g., salbutamol or ipratropium), which relaxes smooth muscles and widens the airways.
Resting tongue posture | 2 weeks
  The resting tongue posture refers to the position of the tongue when the body is at rest, without any active movements such as speaking, chewing, or swallowing. It plays a crucial role in oral and facial development, as well as in maintaining proper function of the airway.
3-Day Food Diary | up to 18 months
  The primary purpose of the 3-Day Food Diary is to accurately record the types and quantities of food and beverages consumed over the course of three consecutive days. It helps to:
  Provide a snapshot of typical eating behaviors and meal patterns.
  Identify potential nutritional deficiencies or imbalances.
  Assess the relationship between diet and health outcomes in clinical studies

CONTACTS AND LOCATIONS:
Overall Officials: Sylwia Mętel, PhD, Study Director — University of Physicsl Culture in Krakow, Poland al. Jana Pawła II 78, 31-571 Kraków
Locations (1):
- Health Resort 'Wieliczka' Salt Mine in Wieliczka, Wieliczka, Wieliczka, Poland

IPD SHARING:
Plan to Share IPD: No